CLINICAL TRIAL: NCT02931344
Title: Biomarkers in Obese Patients With Knee Osteoarthritis Following a Significant Weight Loss
Brief Title: Biomarkers in Obese Patients With Knee Osteoarthritis; Weight Loss
Acronym: BIO-LOSEIT-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henrik Gudbergsen (Other)
Responsible Party: Sponsor-Investigator, Henrik Gudbergsen, MD, PhD, Parker Research Institute
Organization: Parker Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 137.04
Record Dates: First submitted 2016-09-23; First posted 2016-10-13 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Osteoarthrtis; Obesity
Keywords: Osteoarthrtis; Obesity; Liraglutide 3 mg; Liraglutide; Biomarkers
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensive dietary intervention (Experimental): Supervised dietary weight loss program lasting 8 weeks
  Interventions: Dietary Supplement: Dietary Supplement: Dietary Supplement: Intensive dietary intervention

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Dietary Supplement: Intensive dietary intervention — Participants receive a hypo-caloric formula diet containing 800 to 1,000 kcal/day. The formula diet consists of ready-to-use meal bars and powders to mix with water to make shakes, soups, or porridge. The weight loss programme consists of an 8-week period with full meal replacement by a standard liquid energy intake protocol. To facilitate compliance with the programme, participants will be scheduled for weekly facility-based group sessions with 6-8 participants led by a dietician. The recommendations for daily nutrient intake will be met.

SUMMARY:
This is a substudy to a randomised trial investigating the effect of liraglutide on body weight and pain in overweight or obese patients with knee osteoarthritis (NCT02905864).

This substudy aims to investigate any changes in biomarkers associated with the initial 8-week weight loss intervention

DETAILED DESCRIPTION:
In the parent trial, patients will be subjected to an 8-week diet intervention phase including a low-calorie diet and dietetic counselling, after which they will be randomised to receive either liraglutide 3 mg or liraglutide 3 mg placebo as an add-on to dietetic guidance on re-introducing regular foods and a focus on continued motivation to engage in a healthy lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Same as parent trial (NCT02905864)

Exclusion Criteria:

* Same as parent trial (NCT02905864)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in collagen II degradation fragment α-C2M | Week -8 to 0
  Blood sampling

SECONDARY OUTCOMES:
Change in collagen II degradation fragment β-C2M | Week -8 to 0
  Blood sampling
Change in non-coding RNA type snoRNAs U38 and U48 | Week -8 to 0
  Blood sampling
Change in miRNA-454 | Week -8 to 0
  Blood sampling
Change in miRNA let-7e | Week -8 to 0
  Blood sampling
Change in Nesfatin-1 | Week -8 to 0
  Blood sampling

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Frederiksberg, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No